CLINICAL TRIAL: NCT00956293
Title: 6-month, Open-label, Randomized, Multicenter, Prospective, Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Everolimus in de Novo Renal Transplant Recipients Participating in the Eurotransplant Senior Program
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of Everolimus in de Novo Renal Transplant Recipients Participating in the Eurotransplant Senior Program
Acronym: Senator
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated because the required sample size of 240-260 de novo senior renal transplant patients was not achieved within a reasonable time.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE19; EudraCT-NO. 2008-005109-20; 2008-005109-20
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Basiliximab; Mycophenolic Acid; Everolimus; Cyclosporine; Adrenal Cortex Hormones

ARMS (2):
- Control group (Active Comparator): During the pre-randomized treatment phase, all participants received a CNI-based regimen consisting of basiliximab, mycophenolic acid (MPA), cyclosporin A (CsA) and corticosteroids (optional). Upon randomization, participants in this group continued with a CNI-based regimen of MPA and CsA.
  Interventions: Drug: Basiliximab; Drug: Enteric Coated Mycophenolic Acid (MPA); Drug: Cyclosporin A (CsA); Drug: Corticosteroids
- Everolimus group (Experimental): During the pre-randomized treatment phase, all participants received a CNI-based regimen consisting of basiliximab, mycophenolic acid (MPA), cyclosporin A (CsA) and corticosteroids (optional). Upon randomization, participants in this group made a stepwise switch to a CNI-free regimen of everolimus and MPA.
  Interventions: Drug: Basiliximab; Drug: Enteric Coated Mycophenolic Acid (MPA); Drug: RAD001; Drug: Cyclosporin A (CsA); Drug: Corticosteroids

INTERVENTIONS:
Drug: Basiliximab — On day 0, 2 hours prior to transplant and day 4 post-transplant, 20 mg x2 were given to all participants. Post randomization, 20mg at weeks 7 and 12 were given to the Everolimus group.
  Other Names: Simulect
Drug: Enteric Coated Mycophenolic Acid (MPA) — A loading dose regimen of 2880 mg/day during weeks 1 and 2 (pre-randomization) were given. During weeks 3 - 6 (pre-randomization), 2160 mg/day were given and during weeks 7 - 24, 1440 mg/day were given if tolerated. Dose reductions due to side effects were possible.
  Other Names: Myfortic
Drug: RAD001 — Upon randomization, 3 mg (od) on Day 1, and 3 mg (1.5 mg every 12 hours) on Day 2 was given. Afterwards, the dosage was based on blood trough level (5 - 10 ng/mL).
  Other Names: RAD001, Certcian
  Arms: Everolimus group
Drug: Cyclosporin A (CsA) — Dosage was based according to blood level
  Other Names: Sandimmun Optoral
Drug: Corticosteroids — Dosage was administered according to local standards and administration was optional as per clinical need and the Investigators' discretion. Steroid withdrawal occurred after week 2 (pre-randomization).

SUMMARY:
This study wants to address whether a calcineurin-inhibitor (CNI)-free regimen six weeks after transplantation for Eurotransplant Senior Program (ESP) patients is as safe and well tolerated as standard treatment but optimizing immunosuppressive therapy with benefits in renal function, new-onset diabetes mellitus, cardiovascular risk, cancer and allograft nephropathy.

ELIGIBILITY:
Inclusion criteria:

* Patients receiving a primary kidney from a donor aged > 65 years
* In the Eurotransplant Senior Program
* Recipients of de novo cadaveric kidney transplants

Exclusion criteria:

* Multi-organ recipients (e.g., kidney and pancreas)
* Patients receiving a kidney from a non-heart beating donor
* Patients who are recipients of A-B-O incompatible transplants
* Patients with already existing antibodies against the HLA-type of the receiving transplant
* Patients who have received an investigational immunosuppressive drug within four weeks prior to study entry (Baseline visit 1)
* Patients with thrombocytopenia, with an absolute neutrophil count of < 1,500/mm³ or leucopenia or hemoglobin < 6 g/dL
* Patients who are HIV, HCV RNA, or Hepatitis B surface antigen positive
* Evidence of severe liver disease
* Females at randomization who will be not considered post-menopausal

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Koeln-Merheim
  - Novartis Investigative Site, München

REFERENCES:
- [Derived] Brakemeier S, Arns W, Lehner F, Witzke O, Vonend O, Sommerer C, Muhlfeld A, Rath T, Schuhmann R, Zukunft B, Kroeger I, Porstner M, Budde K. Everolimus in de novo kidney transplant recipients participating in the Eurotransplant senior program: Results of a prospective randomized multicenter study (SENATOR). PLoS One. 2019 Sep 19;14(9):e0222730. doi: 10.1371/journal.pone.0222730. eCollection 2019. PMID 31536556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a main period and a 54 month observation follow-up period. The main period included a pre-randomized treatment phase (6 weeks) and a randomized treatment phase (18 weeks). All randomized participants, who participated in the main period, were eligible for the follow-up period.
Pre-assignment Details: At baseline (BL) 1 (pre-randomization), eligible participants received a CNI-based regimen for 6 weeks. At BL2 (randomization), eligible participants were randomized in a 1:2 ratio to the control group or everolimus group.
Groups:
- Pre-randomized Group: Participants, who met BL1 eligibility, were enrolled into the study.
Period: Main Period (Pre-randomization)
Arm/Group | Control Group | Everolimus Group | Pre-randomized Group
Started | 0 | 0 | 207
Enrolled Safety Set | 0 | 0 | 203
Completed | 0 | 0 | 77
Not Completed | 0 | 0 | 130
Not completed — Not specified (data missing) | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Abnormal test procedure result | 0 | 0 | 2
Not completed — Administrative problems | 0 | 0 | 6
Not completed — Graft loss | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 12
Not completed — Lack of Efficacy | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 36
Not completed — Abnormal laboratory value | 0 | 0 | 44
Period: Main Period (Randomization)
Arm/Group | Control Group | Everolimus Group | Pre-randomized Group
Started | 24 | 53 | 0
Full Analysis Set | 24 | 51 (Two participants, randomized to this arm, did not receive everolimus.) | 0
Randomized Safety Set | 24 | 51 | 0
Completed | 23 | 26 | 0
Not Completed | 1 | 27 | 0
Not completed — Abnormal laboratory value | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 10 | 0
Not completed — Adverse Event | 0 | 15 | 0
Period: Follow-up Period
Arm/Group | Control Group | Everolimus Group | Pre-randomized Group
Started | 20 | 32 | 0
Completed | 0 | 0 | 0
Not Completed | 20 | 32 | 0
Not completed — Follow-up period was terminated. | 20 | 32 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Everolimus Group | Total
Number analyzed (Participants) | 24 | 51 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (3.1) | 68.4 (3.3) | 68.7 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 26 | 34
  Male | 16 | 25 | 41

OUTCOME MEASURES:

1. Primary Outcome: Renal Function by Glomerular Filtration Rate (GFR) Via Cockcroft-Gault Method
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Month 6
Population: This outcome measure was not analyzed because a total of 244 completed subjects were needed to have a power of 80% in detecting a significant difference between treatment groups. Due to early termination, the study was limited by a small sample size; hence, the planned analysis was not done.
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Renal Function by GFR Via Modification of Diet in Renal Diseases (MDRD) and Nankivell Method
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Renal Function by Serum Creatinine
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Months 6, 12, 24, 36, 48 and 60
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Biopsy Proven Acute Rejection (BPAR), Graft Loss and Death
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Months 6, 12, 24, 36, 48 and 60
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Occurrence of Treatment Failures
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Evolution of Renal Function (Creatinine Slope)
Description: The study was terminated prematurely and not powered for efficacy.
Time Frame: Week 7, Month 6
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: CD25 Saturation on Lymphocytes
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Experienced Adverse Events, Serious Adverse Events and Death
Description: Participants with adverse events (serious plus non-serious), serious adverse events and death were reported.
Time Frame: Months 6, 12, 24, 36, 48 and 60
Population: Randomized Safety Set: This set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 24 | 51
Participants
  Adverse events (serious and non-serious) | 21 | 50
  Serious adverse events | 11 | 28
  Deaths | 0 | 0

9. Secondary Outcome: Renal Function by GFR Over Time
Time Frame: Months 12, 24, 36, 48 and 60
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Renal Function by Proteinuria
Time Frame: Months12, 24, 36, 48 and 60
Population: as for outcome 1
Arm/Group | Control Group | Everolimus Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Control Goup: During the pre-randomized treatment phase, all participants received a CNI-based regimen consisting of basiliximab, mycophenolic acid (MPA), cyclosporin A (CsA) and corticosteroids (optional). Upon randomization, participants in this group continued with a CNI-based regimen of MPA and CsA.
Arm/Group | Control Goup | Everolimus Group
Serious Adverse Events (participants affected / at risk) | 11/24 | 28/51
Other Adverse Events (participants affected / at risk) | 15/24 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Goup (N=24) | Everolimus Group (N=51)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 3
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
TRANSPLANT REJECTION (Immune system disorders) | 1 | 0
BK VIRUS INFECTION (Infections and infestations) | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 | 1
FEBRILE INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
GENITAL HERPES (Infections and infestations) | 0 | 1
HEPATIC CYST INFECTION (Infections and infestations) | 1 | 0
HERPES ZOSTER OTICUS (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 2 | 1
PNEUMONIA (Infections and infestations) | 2 | 4
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 5
UROSEPSIS (Infections and infestations) | 0 | 1
GRAFT DYSFUNCTION (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 4 | 5
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
FACIAL NERVE DISORDER (Nervous system disorders) | 0 | 1
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 | 1
ANURIA (Renal and urinary disorders) | 1 | 0
NEPHROSCLEROSIS (Renal and urinary disorders) | 1 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 2
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 1
LYMPHOCELE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Goup (N=24) | Everolimus Group (N=51)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 6
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 20
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 9
CONSTIPATION (Gastrointestinal disorders) | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 0 | 10
FLATULENCE (Gastrointestinal disorders) | 0 | 4
NAUSEA (Gastrointestinal disorders) | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 7 | 13
PYREXIA (General disorders) | 4 | 5
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 2 | 4
NASOPHARYNGITIS (Infections and infestations) | 1 | 5
URINARY TRACT INFECTION (Infections and infestations) | 6 | 22
BLOOD CREATININE INCREASED (Investigations) | 1 | 5
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 4
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 12
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 4
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 5
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 3
INSOMNIA (Psychiatric disorders) | 1 | 3
PROTEINURIA (Renal and urinary disorders) | 0 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.